CLINICAL TRIAL: NCT02832713
Title: Randomized Controlled Trial Comparing Botulin Toxin Versus Hyaluronic Acid by Intra-articular Injection for the Treatment of Painful Knee Osteoarthritis
Brief Title: Trial Comparing Botulin Toxin Versus Hyaluronic Acid by Intra-articular Injection for the Treatment of Painful Knee Osteoarthritis
Acronym: GOTOX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6122
Record Dates: First submitted 2016-05-27; First posted 2016-07-14 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Painful Unilateral Femorotibial Knee Osteoarthritis of Any Etiology
Keywords: Knee osteoarthritis; Intra-articular botulinum toxin; Hyaluronic acid; Pain; Function
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-articular injection of botulinum toxin A (Experimental)
  Interventions: Drug: Botulinum toxin A ( BoNT-A)
- Intra-articular injection of hyaluronic acid (Active Comparator)
  Interventions: Device: Hyaluronic acid (HA)

INTERVENTIONS:
Drug: Botulinum toxin A ( BoNT-A) — Intra-articular injection of BoNT-A
  Arms: Intra-articular injection of botulinum toxin A
Device: Hyaluronic acid (HA) — Intra-articular injection of Hyaluronic acid
  Arms: Intra-articular injection of hyaluronic acid

SUMMARY:
In France, osteoarthritis affects about 10 million people and knee osteoarthritis represents 35% of cases. It is thought that more than 2.5 million people older than 65 years have knee osteoarthritis.

Currently, osteoarthritis management is based on three major axes:

1. Non-pharmacological means, such as patient education, loss of weight and physical activity
2. General pharmacological treatments: mainly paracetamol and then schedule II and III painkillers as well as nonsteroidal anti-inflammatory agent.
3. Intra-articular pharmacological treatments:

   1. Intra-articular injections of corticosteroids: they are recommended during hydarthrotic flare-ups
   2. Intra-articular injections of hyaluronic acid (HA) (viscosupplementation) in the absence of intra-articular effusion. However, their efficacy is questioned by most experts in the case of symptomatic knee osteoarthrosis.
4. Sometimes, surgery is the only therapeutic option. However, besides the fact of exposing patients, who are sometimes frail, to several peri- and post-operative complications, the recovery rate (variable according to the prosthesis type and ranging from 5% to 25% at 9 years) in an ageing population justifies waiting as much as possible before surgery. Therefore, it is important to test new therapeutic options for symptomatic osteoarthrosis that will allow postponing the surgical treatment.
5. The use of botulinum toxin (BoNT-A) could thus represents an interesting alternative. BoNT-A is habitually used by intra-muscular injection for its myorelaxant effect in the management of painful reactive periarticular muscle contractures. However, BoNT-A has also antalgic activity independently of the myorelaxant effect. This allows explaining in part the antalgic effect of intra-articular BoNT-A injection. In the literature, six randomized controlled studies (RCS) have compared BoNT-A and intra-articular injections of corticosteroids, hyaluronic acid, or placebo. Only two RCS concerned knee osteoarthritis and compared BoNT-A to corticosteroids and a placebo, respectively, with a significant antalgic effect only in the groups treated with BoNT-A. No study has compared yet the intra-articular injection of BoNT-A to the viscosupplementation by HA in knee osteoarthritis and this is the aim of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Painful, or predominantly unilateral painful, knee osteoarthritis of any etiology
* Knee without clinical signs of intra-articular effusion
* Kellgren score ≥ II on X-ray
* WOMAC pain sub-score ≥ 5 in the month preceding the inclusion visit

Exclusion Criteria:

Clinical:

* Inflammatory arthropathy,infectious, neoplastic within the past year
* Neuromuscular pathology
* Cardiorespiratory pathology or any other severe disease that interferes with the functional capacities
* Any decompensated or unstable chronic pathology
* Glomerular filtration rate (GFR)<15 mL/min/1.73m²) within the past 6 months
* HBA1c in diabetic people > 12% within the past 6 months
* BMI ≥ 35kg/m2
* Infection: joint, general, distant, cutaneous
* Foreign material in the knee to be treated: prosthesis, osteosynthesis material
* Severe coagulation problem: platelets <100000/mm3 within the past 6 months
* Allergy to BoNT-A
* Allergy to HA
* Pregnant or breast-feeding women
* Treatment with aminoglycosides or direct oral anticoagulants
* Treatment with VKA (antihemorrhagic vitamin) if INR (International Normalized Ratio) higher than 3 within the past month
* Change of anti-pain treatment less than 2 weeks before enrolment
* Treatment with III pain killers or corticosteroids because of intense pain that does not respond to schedule I and II pain-killers
* Intra-articular injection of corticosteroids in the previous two months
* Viscosupplementation and/or injection of BoNT-A in the knee to be treated within the past 6 months
* Injection of BoNT-A (except the knee to be treated) within the past 3 months
* Swallowing troubles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of pain measured using the WOMAC pain sub-score | Change from baseline WOMAC pain sub-score at 3 months

SECONDARY OUTCOMES:
Evaluation of the antalgic effect of BoNT-A vs hyaluronic acid measured using a verbal rating scale (VRS) | 1 week after injection
Evaluation of the patients' functional improvement based on the WOMAC score ("stiffness and function sub-score" and total score) | Before injection, 1 month, 3 months and 6 months following injection
Evaluation of the patients' functional improvement using the Timed Up-and-go Test | Before injection, 1 month, 3 months and 6 months following injection
Evaluation of the quality of life based on the SF-36 score | Before injection, 1 month, 3 months and 6 months following injection
Frequency, seriousness and severity of adverse event reactions | during the 6 months following injection
Changes in pain treatment score (using a correspondence table) | Change from baseline pain treatment score at 6 months
Changes in muscular strenght et muscular trophicity (using dynanometer and measure of knee and thin circumference) | Before injection, 1 month, 3 months and 6 months following injection
Changes in passive and active articular knee amplitude, by goniometry | Before injection, 1 month, 3 months and 6 months following injection

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No